CLINICAL TRIAL: NCT01460797
Title: Effects of a Caloric Restriction High/Low-glycemic Index Diets and in Combination With Metformin on Glucose Metabolism, Lipid Profile and Body Composition in Overweight/Obese Subjects
Brief Title: Metabolic Effects of a Caloric Restriction High/Low Glycemic Index Diet Plus Metformin in Overweight/Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caio Eduardo Gonçalves Reis (Other)
Collaborators: University of Brasilia (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fund to support research of the Federal District, Brazil (Unknown)
Responsible Party: Sponsor-Investigator, Caio Eduardo Gonçalves Reis, Sub-Investigator, University of Brasilia
Organization: University of Brasilia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Glycemic index and Metformin
Record Dates: First submitted 2011-10-17; First posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: Glycemic index; Caloric restriction; Energy intake; Glucose; Lipid Metabolism; Cholesterol; HDL Cholesterol; LDL Cholesterol; Obesity; Metformin
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Glycemic Index (Other): Hypocaloric diet with predominating high glycemic index foods
  Interventions: Other: Glycemic Index Diets and Metformin hydrochloride
- Low Glycemic Index (Other): Hypocaloric diet with predominant low glycemic index foods
  Interventions: Other: Glycemic Index Diets and Metformin hydrochloride
- Low Glycemic Index plus Metformin (Other): Hypocaloric diet with predominant low glycemic index foods plus Metformin (1g/d)
  Interventions: Other: Glycemic Index Diets and Metformin hydrochloride

INTERVENTIONS:
Other: Glycemic Index Diets and Metformin hydrochloride — 1g of Metformin hydrochloride a day in High Glycemic Index Diet
  Other Names: High Glycemic Index; Low Glycemic Index; High Glycemic Index plus Metformin

SUMMARY:
The prevalence of obesity and Type 2 diabetes has increased dramatically worldwide. Research on Glycemic Index (GI) diets has been largely developed, however the combination with metformin in humans was not investigated yet. We hypothesized that the low-GI diet in combination with metformin would elicit greater improvements on glucose metabolism, lipid profile and body composition on overweight or obese type 1 subjects. This study aims to evaluate the metabolic effects of the adoption of dietary advice to follow caloric restriction high/low GI diets, and low-GI diet associated with metformin on glucose metabolism, lipid profile and body composition on overweight or obese type 1 subjects.

DETAILED DESCRIPTION:
All groups (Low/High-GI and Low-GI + Metformin) showed significant reduction in anthropometric parameters, but only Low-GI and Low-GI + Metformin groups have an improvement in body composition parameters. In addition, the Low-GI group achieved better results in metabolism of carbohydrates (glucose, insulin, Cederholm Index, and HOMA-β) and lipids (Chol, TAG, LDL-C, VLDL-C, and TC/HDL-c). These results show the benefits of Low-GI diet on metabolic parameters in overweight or obese type 1 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Participants were adults (18-50 y), with body mass index (BMI) between 25-35 kg/m².
* Subjects with adequate glycemic and insulinemic response after oral glucose tolerance test: Hypocaloric diet with predominating high glycemic index foods;
* Subjects with altered glycemic response presented at the 120 min point either glycemia <140mg/dL and insulin level >40 µUI/ml: Hypocaloric diet with predominant low glycemic index foods;
* Subjects with impaired glucose tolerance presented at the 120 min point glycemia 140 - 199mg/dL and insulin >40 µUI/ml: Hypocaloric diet with predominant low glycemic index foods and metformin.

Exclusion Criteria:

* Smokers
* Pregnant or lactating
* Diagnosis of any metabolic diseases
* Were under medication and therapeutic diet, except oral contraceptive for women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolism | 0 and 4 months
  2-hour oral glucose tolerance test (Glucose and Insulin levels), glucose and insulin IAUC, HbA1c, HOMA-IR, HOMA-β, and Cederholm Index.

SECONDARY OUTCOMES:
Lipid Profile | 0 and 4 months
  Cholesterol, TAG, LDL-C, VLDL-C, HDL-c, and Cholesterol/HDL-c ratio
Body Composition | 0 and 4 months
  Body weight, Height, Body mass index, Body fat mass, Free fat body mass, Waist circumference.
Clinical Assessment | 0 and 4 months
  FSH hormone, urea, creatinine, and uric acid urinary levels
Food Intake | 0 and 4 months
  Energy intake, macronutrients and fiber consumption

CONTACTS AND LOCATIONS:
Overall Officials: Teresa HM da Costa, Ph.D., Study Director — University of Brasilia
Locations (1):
- School of Health Sciences, University of Brasília, Brasília, Federal District, Brazil